CLINICAL TRIAL: NCT04390607
Title: A Research Study to Determine if a Leukocyte Esterase Electrochemical Assay Can be Used as a Marker for Periprosthetic Joint Infection
Brief Title: Leukocyte Esterase Sensor Test
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: 2020Cleu
Record Dates: First submitted 2020-05-11; First posted 2020-05-15 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Prosthetic Joint Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects undergoing revision joint surgery
  Interventions: Diagnostic Test: leukocyte esterase electrochemical assay

INTERVENTIONS:
Diagnostic Test: leukocyte esterase electrochemical assay — A sample of blood drawn for routine standard of care laboratory assessments will be used to also test the new electrochemical assay. This is a validation study and the results of the electrochemical assay will not be used to treat patients

SUMMARY:
The primary objective of this study is to assess the diagnostic efficacy of the quantitative electrochemical LE biosensor for periprosthetic joint infection (PJI). The secondary objective of this study is to assess the utility of d-lactase as adjunct biomarker to LE in making a diagnosis of PJI.

ELIGIBILITY:
Inclusion Criteria:

1: consecutive patients undergoing at least one of the following procedures: presumed aseptic revision arthroplasty, irrigation and debridement, radical resection for periprosthetic joint infection

Exclusion Criteria:

1. known active gout flare
2. existing corrosion or metallosis
3. inflammatory arthritis
4. preexisting diagnosis of infection in the same joint
5. patients undergoing second-stage procedure for infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a prospective study with consecutive revision joint surgery patients determined to be in one of three groups: 1) patients undergoing revision joint replacement for presumed aseptic loosening, 2) patients undergoing irrigation and debridement with implant retention, and 3) patients undergoing two stage revision for infection. We will also recruit a small number of patients undergoing primary joint replacement (Jefferson hospital only).
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Receiver Operating Curve (ROC) analysis | 20 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Langone Health, New York, New York, United States